CLINICAL TRIAL: NCT04446442
Title: Biologic Effects and Efficacy of Cerebellar tDCS in Children With Autism Spectrum Disorder
Brief Title: Cerebellar tDCS in Children With Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Peter Tsai, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: UTSW 022017-071; W81XWH1910249 (Other Grant/Funding Number: US DEPARTMENT OF DEFENSE)
Record Dates: First submitted 2019-11-12; First posted 2020-06-25 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Full Administration of Transcranial Direct Current Stimulation (Experimental): Each subject will undergo psychosocial and behavioral assessments at a session prior to the administration of tDCS. The second session will include the tDCS Administration; a current of 1 mA will be administered over 20 minutes to the right crusI/II area of the cerebellum with a 15 second fade in period at the beginning and a 15 second fade out period at the end. During the tDCS administration, subjects will undergo functional MRI scanning. After the tDCS administration, subjects will repeat psychosocial and behavioral assessments.
  Interventions: Device: tDCS
- Sham Administration of Transcranial Direct Current Stimulation (Sham Comparator): Each subject will undergo psychosocial and behavioral assessments at a session prior to the administration of tDCS. The second session will include the tDCS Administration; a current of 1mA increased over 15 seconds and immediately decreased over 15 seconds to provide sensation associated with tDCS. During the sham administration, subjects will undergo functional MRI scanning. After the tDCS administration, subjects will repeat psychosocial and behavioral assessments.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — A current of 1 mA will be administered for 20 minutes of with either anodal or cathodal tDCS administration to the right crus I/II area of the cerebellum.

SUMMARY:
The purpose of this research study is to investigate whether tDCS to the cerebellum (specifically, the right crus I/II area of the cerebellum) of children and young adults with autism spectrum disorders (ASD) is safe and to examine its effects on some of the symptoms of ASD, such as repetitive behaviors and hyperactivity.

DETAILED DESCRIPTION:
The study will be randomized, double-blind, and controlled. It will involve a group of 60 children with ASD (diagnosed with the Autism Diagnostic Observation Schedule (ADOS-2) by a research-reliable clinician) coming in for an orientation day, where participants will be acclimated to the testing environment, as well as undergo safety screening, and a mock MRI. The investigators will recruit from a sample of children diagnosed with ASD (The diagnosis must be made by experienced, research reliable clinicians using gold standard measures including the Autism Diagnostic Observation schedule Second Edition Study, or ADOS-2 and a diagnostic and developmental parent interview). The investigators will request this information from the institution where the diagnosis was given with parent/caregiver permission. Diagnostic information will be reviewed by the study neuropsychologist, and if additional testing is needed to update or confirm the diagnosis, the investigators will administer an ADOS-2 here at UTSW prior to other baseline measures. If diagnostic information from a previous CADD clinic visit or an outside institution by a research reliable clinician is current, the investigators will accept it.

Participants will complete in a variety of tasks during a pre-treatment visit. In addition, baseline behavioral measurements will be performed. These tests include an abbreviated measure of cognitive ability using the Stanford Binet-Fifth Edition, interpretation of facial expressions, memory for faces, reading the mind in the eyes, triangle animations, cyberball /social ball throwing, dimensional card change sort, and caregiver-completed behavioral scale including the Autsim Spectrum Rating Scale (ASRS). Participants will also be asked about their mood before, during, and after treatment. Participants will then be randomly assigned into either a sham treatment group or an active treatment group. The next time the participants come in, participants vitals will be monitored in addition to eye monitoring and will undergo either 1 mA for 20 minutes of anodal or cathodal tDCS administration to Right Crus I/II area of the cerebellum or sham treatment. Participants will undergo fMRI imaging prior, during, and after anodal or cathodal tDCS. After the scans, testing will be repeated and include interpretation of facial expression, memory for faces, reading the mind in the eyes, triangle animations, theory of mind, cyberball/social ball throwing, and dimensional card change sort. At the end of the visit parents/guardians/participants will receive a safety questionnaire asking about the presence and severity of the possible side effects. The participants will then follow up in 1 week with the safety questionnaire and at 1 month with the safety questionnaire and the Autism Spectrum Rating Scale.

Study Procedures:

Investigators, including those involved in questionnaire and behavioral scales administration and fMRI scanning/interpreting will be blinded to which treatment group participants are in. Staff members in charge of applying tDCS will be aware of what treatment group the participant is in but will not be involved in analysis of data to ensure blinding of results. As far as the tDCS procedure goes, the device consists of a programmable current source with a rechargeable battery with two wires connected to electrodes in fabric pads. The device cannot be plugged into an outlet while the electrodes are connected, ensuring safety. tDCS pads are moistened with 0.9% normal saline and placed on the participant's scalp using elastic bands. During stimulation, the electrodes will apply 1 mA of constant DC electrical current. Current will be increased over 10-60 seconds. The current will be applied for no more than 20 minutes, after which the current is decreased over 10-60 seconds. In sham tDCS, the current is increased and then immediately decreased to provide sensations associated with tDCS (mild tingling or itching, which blinds the participant).

Testing will take place before (on orientation day) and after tDCS. Baseline testing includes an ADOS-2 if deemed necessary, an abbreviated cognitive measure, interpretation of facial expressions, memory for faces, reading the mind in the eyes, triangle animations, cyberball /social ball throwing, dimensional card change sort, and caregiver-completed behavioral scale including the Autsim Spectrum Rating Scale.. Testing immediately after tDCS includes only the following: interpretation of facial expressions, memory for faces, reading the mind in the eyes, triangle animations, theory of mind, cyberball/social ball throwing, and dimensional card change sort.

Participants with ASD will come in on designated orientation days and be assigned an alphanumeric identifier to ensure confidentiality. An initial safety screening will be done to ensure no exclusion criteria are met. Participants will then be randomly split into either a sham group or a treatment group. Baseline testing will be completed. Participants will then be allowed to explore and become acclimated with study equipment, and a mock MRI will be done on the first visit at the UTSW Advanced Imaging Research Center (AIRC).

Participants will be desensitized to the sounds and tactile sensations of the fMRI environment while in a space similar to that of the scanner bore. Participants will practice remaining still within the mock MRI while viewing a movie, and biofeedback is used to train participants to keep their movement <1mm during practice periods of 10 minutes. Participants should be able to complete all of the screening in one visit. If participants cannot due to time constraints participants will be brought back in on a different day to complete the screening visit.

The next time participants return, participants will be hooked up to vitals and eye movement monitoring and will be placed in the fMRI machine so the "before" scanning can begin. After this "before" scan, tDCS electrodes will be applied and participants will again be placed in the fMRI machine for the "during" scan. As soon as scanning begins, tDCS (either sham or treatment of 1 mA for 20 minutes of anodal tDCS administration to the Right Crus I/II area of the cerebellum) will begin as well. During tDCS treatment caregivers will receive a safety questionnaire for them to assess any side effects occurring in their child. After this scan, the tDCS electrode will be removed, and a final "after" fMRI scan will take place. The safety questionnaire will be given after tDCS at the end of the visit and behavioral tests are complete.The time estimated for all of this is about 90-180 minutes.

The Safety Questionnaire will be assessed again with follow-up visits 1 week and 1 month afterwards using the same caregiver-completed scales.

ELIGIBILITY:
Inclusion Criteria:

* 4-17 years old
* Diagnosed with ASD and ADOS-2
* IQ Score no less than 70 (1.5 Standard Deviations below the mean)
* Language Level (Speech consists of, at minimum, flexible, spontaneous, simple, sentences)

Exclusion Criteria:

* Brain implants, metal implants, pacemakers, or biomedical devices
* Diagnosis of epilepsy
* Hearing or visual impairments
* History of brain injury
* Known brain abnormalities not associated with ASD

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-06-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of tDCS associated side effects assessed by tDCS Safety Assessment | Post-Intervention up to one month
  Observe whether tDCS to the cerebellum (specifically, the right crus I/II area of the cerebellum) of children and young adults diagnosed with autism spectrum disorders (ASD) is safe and easily tolerated using a tDCS Safety Assessment

SECONDARY OUTCOMES:
Change in Autism Spectrum Disorder Symptoms assessed by NEPSY-2 Subtests | Pre-Intervention at 1 week and Post-Intervention at 1 hour
  Observe tDCS to the cerebellum (specifically, the right crus I/II area of the cerebellum) of children and young adults diagnosed with autism spectrum disorders (ASD) and its effects on some of the symptoms of ASD, related to social behavior and cognition. The NEPSY-2 subtests include: Memory for Faces, Theory of Mind, and Affect Recognition. The NEPSY-2 subtests are designed to assess abilities related to memory, learning, and social perception.
Change in Autism Spectrum Disorder Symptoms assessed by Reading the Mind in the Eyes | Pre-Intervention at 1 week and Post-Intervention at 1 hour
  Observe tDCS to the cerebellum (specifically, the right crus I/II area of the cerebellum) of children and young adults diagnosed with autism spectrum disorders (ASD) and its effects on some of the symptoms of ASD, related to social behavior and cognition. This will be assessed by Reading the Mind in the Eyes, a measure of complex mental state recognition.
Change in Autism Spectrum Disorder Symptoms assessed by Triangle Animations/Social Perception Task | Pre-Intervention at 1 week and Post-Intervention at 1 hour
  Observe tDCS to the cerebellum (specifically, the right crus I/II area of the cerebellum) of children and young adults diagnosed with autism spectrum disorders (ASD) and its effects on some of the symptoms of ASD, related to social behavior and cognition. The Triangle Animations/ Social Perception Task assesses Theory of Mind mental functions such as belief and intention.
Change in Autism Spectrum Disorder Symptoms assessed by Cyberball/Social Ball Throwing Task | Pre-Intervention at 1 week and Post-Intervention at 1 hour
  Observe tDCS to the cerebellum (specifically, the right crus I/II area of the cerebellum) of children and young adults diagnosed with autism spectrum disorders (ASD) and its effects on some of the symptoms of ASD, related to social behavior. The Cyberball/Social Ball Throwing Task assesses engagement in social interaction.
Change in Autism Spectrum Disorder Symptoms assessed by Dimensional Change Card Sort | Pre-Intervention at 1 week and Post-Intervention at 1 hour
  Observe tDCS to the cerebellum (specifically, the right crus I/II area of the cerebellum) of children and young adults diagnosed with autism spectrum disorders (ASD) and its effects on some of the symptoms of ASD, related to cognition. The Dimensional Change Card Sort is a measure of cognitive flexibility, also known as task switching or set shifting.
Change in Autism Spectrum Disorder Symptoms assessed by Autism Spectrum Rating Scale | Pre-Intervention at 1 week and Post-Intervention at 1 week and 1 month
  Observe tDCS to the cerebellum (specifically, the right crus I/II area of the cerebellum) of children and young adults diagnosed with autism spectrum disorders (ASD) and its effects on some of the symptoms of ASD, such as repetitive behaviors and hyperactivity. The Autism Spectrum Rating Scale (ASRS) is a nationally-standardized, norm-referenced checklist designed to identify symptoms, behaviors, and associated features of Autism Spectrum Disorders in children and adolescents. Using a five-point Likert rating scale (1- Never, 2- Rarely, 3- Occasionally, 4- Frequently, 5- Very Frequently), parents/caregivers are asked to evaluate how often they observed specific behaviors in the child or adolescent in areas such as socialization, communication, unusual behaviors, behavioral rigidity, sensory sensitivity, and self-regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Tsai, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Children's Medical Center, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No